CLINICAL TRIAL: NCT04144764
Title: Quantification of Upper Trapezius Muscle Stiffness Using Supersonic Shear Wave Imaging: Efficacy of Workplace-based Exercise Programme to Reduce Neck and Shoulder Disorders in Working Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEONG Hio Teng, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.269
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Neck Pain; Shoulder Pain
Keywords: upper trapezius; muscle stiffness
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workplace-based exercise group (Experimental)
  Interventions: Other: Workplace-based exercise
- Control group (Sham Comparator)
  Interventions: Other: Ergonomic advice and education

INTERVENTIONS:
Other: Workplace-based exercise — Participants will have to perform 10-week of workplace-based exercise programme which consist of 5 sessions of 10 minutes per week. The workplace-based exercise programme will consist of general stretching and strengthening exercise using resistance tubing for both the neck and upper limb. Specific rotator cuff and scapular muscles strengthening exercise were also included to enhance glenohumeral and scapular kinematics (Appendix). Each participant will receive a set of elastic resistance tubing that comprise red (2kg), green (3kg) and blue (4kg). The exercise programme will be taught by physiotherapist during their baseline assessment. They will be asked to train at the workplace during workdays (Monday to Friday), five times a week during the 10-week intervention. The program built on the principle of progressive overload.
  Arms: Workplace-based exercise group
Other: Ergonomic advice and education — Participants will receive ergonomic training and education on how to adjust their workstations to reduce the ergonomic risk factors when using computers.
  Arms: Control group

SUMMARY:
Objectives: (1) To examine the upper trapezius muscle stiffness using SSI in workers with and without neck/shoulder disorders; and (2) to develop a workplace-based exercise programme to reduce upper trapezius muscle stiffness and to enhance shoulder function and work ability in the working population.

Hypotheses to be tested: (1) Workers with neck/shoulder disorders demonstrate increase upper trapezius muscle stiffness when compared to healthy control; and a cutoff value of the upper trapezius stiffness was established for early identification of individuals at risk of having neck/shoulder disorders in the working population; (2) Workplace-based exercise programme can reduce upper trapezius muscle stiffness and enhance shoulder function and work ability in the working population.

Design: Part A study: Cross-sectional study; Part B study: randomized controlled trial

Subjects: One-hundred office computer workers with or without neck/shoulder pain

Study instruments: Supersonic shear wave imaging

Main outcome measures: Upper trapezius muscle stiffness, Shoulder Pain and Disability Index (SPADI), Neck Disability Index, Disability of the Arm, Shoulder and Hand (DASH), work ability index (WAI).

Data analysis: Between-group comparisons to show differences in the outcome measures will be analyzed using Independent t-test. To compare the treatment effects, repeated-measures analysis of variance test (between-group factor: intervention vs control; within-subject factor: time (baseline, 6 week and 1 year)).

Expected results: Workers with neck/shoulder disorders demonstrate increase upper trapezius muscle stiffness when compared to healthy control. Workplace-based exercise programme can reduce upper trapezius muscle stiffness and enhance shoulder function and work ability in the working population.

ELIGIBILITY:
Inclusion Criteria:

* Office computer workers who worked for a minimum of four hours per day using a computer
* With or without neck/shoulder pian

Exclusion Criteria:

* Involved regular strength training of the neck/upper extremities within the past 12 months;
* history of whiplash, neck/upper limb fractures, previous surgery and previous clinical treatment for a neck/upper limb injury within the last 12 months;
* Fibromyalgia;
* Pregnancy;
* Neurological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-09 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Upper trapezius muscle stiffness | 0, 10-weeks and 1-year
  Supersonic shear wave imaging of the upper trapezius muscles

SECONDARY OUTCOMES:
Change in Shoulder Pain and Disability Score | 0, 10-weeks and 1-year
  The Chinese Version of the Shoulder Pain and Disability Index (SPADI) questionnaire is a validated self-administered questionnaire to evaluate the shoulder pain and disability scores. The questionnaire consists of 13 items with 2 subscales: pain (5 items) and disability (8 items); and the total final score that range from 0 to 100, with higher scores indicate more disability.
Change in Functional score | 0, 10-weeks and 1-year
  The Chinese Version of the Neck Disability Index and Disability of the Arm, Shoulder and Hand (DASH-HKPWH) questionnaire are reliable and validated self-administered questionnaire to evaluate the neck and upper extremity function. The total score is divided by number of answered questions, subtracted 1 and multiplied by 25, in a scale score that range from 0 to 100, with higher scale scores indicate more disability.
Change in Work ability | 0, 10-weeks and 1-year
  The work ability index (WAI) questionnaire will be used to evaluate the work ability. It composes of 7 items that evaluate: 1) current work ability compared with lifetime best; 2) work ability in relation to job demand; 3) number of current diagnosed disorders; 4) estimated work impairment due to disease; 5) sick leave during the past 12 months; 6) own prognosis of work ability; and 7) mental capacities. The score ranged between 7 to 49, with higher scores indicate better work ability.

CONTACTS AND LOCATIONS:
Locations (1):
- CUHK-ORT Sports Injury Research Laboratory, Hong Kong, Hong Kong